CLINICAL TRIAL: NCT04284709
Title: Novel Mat Exergaming to Improve the Physical Performance, Cognitive Function, and Dual-task Walking and Decrease the Fall Risk of Community-dwelling Older Adults
Brief Title: Exergaming for Community-Dwelling Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, CY Song, Prof, National Taipei University of Nursing and Health Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 18-116-B
Record Dates: First submitted 2020-02-20; First posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Elderly; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise group (Experimental): exergames with simultaneous cognitive-physical training
  Interventions: Other: cognitive-physical training
- control group (Active Comparator): multicomponent exercise intervention focused on physical and cognitive training
  Interventions: Other: cognitive-physical training

INTERVENTIONS:
Other: cognitive-physical training — combined physical and cognitive training

SUMMARY:
This study aimed to utilize an interactive exergame mat system to develop a novel cognitive-physical training program and explore the training effects on physical performance, cognitive function, dual-task walking (DTW), and fall risk compared to the control condition.

DETAILED DESCRIPTION:
The exercise group performed exergames with simultaneous cognitive-physical training, while the control group underwent a multicomponent exercise intervention focused on physical and cognitive training. A 2-hour training session was completed weekly for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* aged 65 years or older, and being able to walk independently without any assistive devices

Exclusion Criteria:

* had severe lower-extremity joint pain, cognitive impairment, or visual problems that impeded their participation

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
change in lower-limb muscle strength | before and after 3-month exercise training interventions
  30-second chair stand test
change in upper-limb muscle strength | before and after 3-month exercise training interventions
  30-second arm curl test
change in aerobic endurance | before and after 3-month exercise training interventions
  2-minute step test
change in lower-body flexibility | before and after 3-month exercise training interventions
  chair sit and reach test
change in upper-body flexibility | before and after 3-month exercise training interventions
  back scratch test
change in dynamic balance | before and after 3-month exercise training interventions
  8-foot up and go test
change in static balance | before and after 3-month exercise training interventions
  single-leg stand test
change in grasp strength | before and after 3-month exercise training interventions
  hand grip strength
change in lower limb motor function | before and after 3-month exercise training interventions
  foot tapping test
change in cognitive function | before and after 3-month exercise training interventions
  Montreal Cognitive Assessment
change in cognitive dual-task walking | before and after 3-month exercise training interventions
  8-foot up and go walking while counting
change in motor dual-task walking | before and after 3-month exercise training interventions
  8-foot up and go walking while carrying a tray
change in fall risk | before and after 3-month exercise training interventions
  fall risk questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Yi Song, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- National Taipei University of Nursing and Health Sciences, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided